CLINICAL TRIAL: NCT06060184
Title: Initiative for Clinical Long-read Sequencing - Towards Implementation of Long-read Genome Sequencing in Routine Diagnostics
Brief Title: Initiative for Clinical Long-read Sequencing
Acronym: IonGER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: RWTH Aachen University (Other); Medical University of Hannover (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IonGER
Record Dates: First submitted 2023-09-13; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Genetic Predisposition
Keywords: Long-read sequencing; Rare diseases; Cancer preposition; Translate-NAMSE; German initiative for genomic medicine (genomDE)
MeSH Terms: conditions — Genetic Predisposition to Disease; Rare Diseases | interventions — High-Throughput Nucleotide Sequencing

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retrospective cohort (Experimental): Subjects with unclear molecular cause of the disease. The subjects are clinically characterized in the context of outpatient/ inpatient standard care at the University Hospital Tübingen (UKT) or cooperating locations.
  Interventions: Genetic: Next-Generation Sequencing (NGS)
- Prospective cohort (Experimental): Subjects with indication for genome diagnostics (e.g. within the initiative for genomic medicine (genomDE) based on §64e German Social Code (SGB) Fifth Book (V) (SGB V).
  Interventions: Genetic: Next-Generation Sequencing (NGS)

INTERVENTIONS:
Genetic: Next-Generation Sequencing (NGS) — Sequencing of genomes (Long read NGS)

SUMMARY:
The study aims to comprehensively introduce Long-read Genome sequencing (LR-GS) based genetic testing into clinical routine. In order to demonstrate the superiority of untargeted LR-GS over Short-read Genome sequencing (SR-GS) to establish firm genetic diagnoses, the investigators will rely on a multi-center "Translate Nationale Aktionsbündnis für Menschen mit Seltenen Erkrankungen" (Translate National Action Alliance for People with Rare Diseases Germany, TNAMSE) cohort of unsolved patients with neurological, neurodevelopmental, and imprinting disorders that is expectedly enriched for complex genomic variation. Within the framework of genomDE, the investigators will then implement, for the first time, LR-GS in the diagnostic work-up of a prospective cohort of patients with a broad range of clinical indications including rare diseases and cancer predisposition.

DETAILED DESCRIPTION:
The proposed study aims to develop a blueprint for the implementation of LR-GS in clinical diagnostics. Hence Standard Operating Procedures (SOPs) and guidelines for library preparation, bioinformatic analysis, and clinical interpretation will be compiled. Furthermore, the investigators intend to develop an open source 'gold standard' bioinformatics pipeline, addressing all relevant types of genomic alterations, thus providing the bioinformatic basis for a streamlined implementation of LR-GS at other sites. In addition to in-depth phenotype information the availability of SR-GS will be instrumental to benchmark the ability to detect different types of genomic variation. Additional relevant issues for genetic testing such as variant calling in difficult-to-map genomic regions, detection of genomic methylation patterns, characterization of repeat expansion and duplicated genes, and haplotype-phased genome de novo assembly will be addressed. Moreover, based on the strong background in Artificial Intelligence (AI) driven variant prioritization in the consortium, the investigators aim to implement and/or develop tools that enable an efficient prioritization of disease-causing variants. Beyond the usage within the context of the proposed study, generated datasets will be made available according to the Findable, Accessible, Interoperable and Reusable (FAIR) principles for national (German Human Genome-Phenome Archive, GHGA) and international (European Genome-Phenome Archive, EGA, Genome-Phenome Analysis Platform, GPaP) data repositories. the investigators aim to establish a population scale reference dataset for Structural variants (SV), which is absolutely mandatory in the context of rare disease diagnostics.

ELIGIBILITY:
Inclusion Criteria:

* Unclear molecular cause of the disease (retrospective cohort)
* Indication for genome diagnostics (prospective cohort; e.g. within the initiative for genomic medicine (genomDE) based on §64e SGB V)
* Suspected genetic cause of the disease

Exclusion Criteria:

- Missing informed consent of the patient or legal guardian

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Rare Disease (RD) or cancer predisposition syndromes with confirmed diagnosis by LR-GS compared to previous diagnostic methods including SR-GS | Day 1
  A molecular diagnosis is considered confirmed when likely pathogenic or pathogenic variants are identified according to the American College of Medical Genetics and Genomics (ACMG). classification.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Haack, Dr. med., Principal Investigator — University Hospital Tübingen
Locations (1):
- University Hospital Tübingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Yes
The IonGER study will provide data in a pseudonymised manner to national and international databases set up to increase the diagnostic yield through advanced analysis tools and matchmaking against other cohorts
Supporting Information: Analytic Code
Time Frame: Data will become available after analysis and unlimited.